CLINICAL TRIAL: NCT04342936
Title: A Randomized,Open-label Phase III Study of Camrelizumab (SHR-1210) vs. Investigator's Choice of Chemotherapy in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma (cHL)
Brief Title: Study of Camrelizumab (SHR-1210) vs. Chemotherapy in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-317
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-04

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab for Injection (Experimental): Participants receive Camrelizumab 200mg intravenously (IV) on Day 1 of each 2-week cycle
  Interventions: Drug: Camrelizumab
- Chemotherapy (Active Comparator): Participants receive investigator's choice of chemotherapy (Gemox, IGEV or DHAP) for up to 6 cycles.
  Interventions: Drug: Investigator's choice of Chemotherapy

INTERVENTIONS:
Drug: Camrelizumab — A humanized monoclonal immunoglobulin
  Other Names: SHR-1210
  Arms: Camrelizumab for Injection
Drug: Investigator's choice of Chemotherapy — Participants will receive one of the following chemotherapies for up to 6 cycles:
  Gemox: Gemcitabine and Oxaliplatin； IGEV: Ifosfamide, Gemcitabine, Vinorelbine, and Prednisolone； DHAP: Dexamethasone, high-dose Cytarabine (Ara-C) and Cisplatin.
  Arms: Chemotherapy

SUMMARY:
This is an open-label, multicenter, randomized, phase3 trial to evaluate the efficacy of Camrelizumab in patients with relapsed or refractory classic Hodgkin's lymphoma. Participants will be randomized to receive either Camrelizumab monotherapy or chemotherapy of investigators' choice.

The primary hypotheses of this study are that treatment with Camrelizumab prolongs Progression-free Survival (PFS) in participants with relapsed or refractory Classical Hodgkin Lymphoma compared to treatment with Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* With histologically confirmed classic Hodgkin's lymphoma ;
* Relapsed or refractory cHL meet either of the following criteria:

  1. Did not achieve remission or progressed after autologous hematopoietic stem cell transplantation.
  2. Received at least 2 lines of systemic chemotherapy, failed to achieve remission or progressed after the most recent chemotherapy.
* Have measurable disease according to Lugano 2014 criteria
* Eastern Cooperative Oncology Group (ECOG) performance scale of 0 or 1;
* Life expectancy ≥ 12 weeks;
* Has adequate organ function;
* Women of childbearing potential（WOCBP） must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 60 days after the last dose of study treatment. Women of childbearing potential with pregnancy test negative within 7days before entering the group and not in in lactation. Male subjects with WOCBP partner should receive Surgical sterilization or consent to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 120 days after receiving the last dose of study treatment.
* Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

* Active, known or suspected autoimmune disease. Subjects who were in a stable state, do not need systemic immunosuppressive therapy were allowed to participate.
* Concurrent medical condition requiring the use of immunosuppressive medications or glucocorticoids exceeds a daily dose of 10mg prednisone or equivalent within 14 days before drug administration. Topical use of glucocorticoids is allowed.
* Received anti-tumor vaccines or other anti-tumor therapy with immune stimulatory effects within 3 months before the first dose SHR-1210.
* Prior exposure to any PD-1/PD-L1/PD -L 2 or CTLA -4 antibody .
* Participating in other clinical studies or less than 4 weeks by the end of the most recent clinical trial participation;
* Known or suspected interstitial pneumonia;
* Concurrent or history of other malignancies. (Except for patients with skin basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma or cervical carcinoma who received radical treatment and did not relapse in 5 years since treatment initiation).
* Received chemotherapy, radiotherapy,immunotherapy, including topical therapy within 4 weeks. Previous anti-tumor therapy related adverse reactions (except hair loss) did not recover to CTCAE ≤1.
* Prior allo-HSCT.
* ASCT within 90 days.
* Impact of major surgery or severe trauma had been eliminated for less than 14 days.
* Active pulmonary tuberculosis.
* Severe acute or chronic infection requiring systemic therapy.
* Suffering from heart failure (New York Heart Association standard III and given appropriate medical treatment.Uncontrolled coronary artery disease and arrhythmia. History of myocardial infarction within 6 months.
* Live vaccine within 4 weeks before the first dose SHR-1210.Inactivated vaccines against seasonal influenza is allowed.Live attenuated influenza vaccines were not approved for intranasal administration.
* HIV test(s) positive or known AIDS.
* Untreated active hepatitis; Hepatitis B and hepatitis C infection in common.
* Other factors that may lead to the study termination, such as severe disease or abnormal laboratory tests or family or social factors affecting subjects safety or test data and sample collection .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | anticipated 16 months
  Time from randomisation to radiologically confirmed progressive disease

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No